CLINICAL TRIAL: NCT01351493
Title: A Randomized, Double-blind, Placebo-controlled Study on the Safety and Efficacy of Nitric Oxide Gel in Subjects With Pressure Sore
Brief Title: Study on the Safety and Efficacy of Nitric Oxide Gel in Subjects With Pressure Sore
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMR100-IRB-030
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Pressure Ulcer
Keywords: pressure sore; nitric oxide
MeSH Terms: conditions — Pressure Ulcer | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitric oxide gel (Active Comparator)
  Interventions: Drug: Nitric Oxide
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Nitric Oxide — Nitric Oxide Gel, once or twice per day, 12weeks
  Arms: Nitric oxide gel
Drug: placebo — placebo Gel, once or twice per day, 12weeks
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of nitric oxide gel for pressure sore recovery.

DETAILED DESCRIPTION:
Pressure sore is a common problem for patient with bed-ridden. The care of pressure sore cost many social and medical resource, and also effect the quality of life of patients. Current principles of treatment of pressure sore include adequate pain control, optimizing nutritional status, pressure relief, wound cleaning and dressing, infection control and surgical intervention if needed. Wound dressings should be based on wound characteristics. However, for improving wound healing, different dressing materials were developed.

There are increased evidences implicate nitric oxide (NO) synthesis plays an important role in the process of wound healing. Nitric oxide involve in angiogenesis, mediating inflammatory process, cell proliferation and collagen disposition, then improving wound healing. One study used topic NO-gel to mice with second degree burn wound, and found that the NO gel had the potential to enhance burn wound healing by regulation of many cellular processes in the skin. Based on the findings, the investigators hypothesize that NO gel could be used as an alternative method for pressure sore dressing to enhance wound healing.

This is a 12-week study. The investigators plan to enroll 40 subjects. The run-in period is set for screening based on inclusion and exclusion criteria. Baseline data including demographic profiles, medical history and current medications will be obtained, followed by an intact pressure sore inspection. Pressure ulcer stage (developed by NPAUP) , Pressure Ulcer Scale for Healing(PUSH) and Pressure Sore Status Tool(PSST) will be recorded before randomization. Baseline photograph of pressure sore will be taken .

During the treatment phase, a NO gel or placebo gel will be administered on the pressure sore wound by caregiver once or twice daily (decided by doctor according to clinical condition) after standard wound cleaning with normal saline. During the treatment period, the study subjects will be followed- up every 2 weeks to record the wound condition and any side effect. The investigators will use stage, PUSH and PSST, and take serial photograph to monitor wound condition.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who live in nursing home
* Clinical diagnosis of pressure sore > grade II(grade developed by NPAUP)
* without acute illness required hospitalization
* able to understanding and signed the Inform Consent Form after detailed description of the treatment and potential risks and benefits

Exclusion Criteria:

* diagnosis of cancer and still on active therapies
* on other medications with pharmacological actions may lead to excessive formation of nitric oxide, or may accentuate drug effects due to excessive formation of nitric oxide
* with systemic infection and need systemic antibiotics
* pressure sore local infection and need topic antibiotic(for pressure sore wound)
* with any known allergic reaction to any ingredient in the 2 gel prescriptions
* Subjects who have been enrolled into any other clinical study in the preceding 3 months prior to randomization

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Pressure ulcer stage assessment after the endpoint of intervention period | 12 weeks

SECONDARY OUTCOMES:
The secondary efficacy end point will be pressure sore scale assessment of improvement. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Shong Liu, M.D., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taichung, Taiwan